CLINICAL TRIAL: NCT03843138
Title: Feasibility and Performance of a Novel 3D Virtual Treatment Planning Software: an International, Multi-centric, Prospective Study
Acronym: 3D IPSCD-TIM
Status: Completed | Type: Observational
Sponsor: AZ Sint-Jan AV (Other)
Collaborators: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other); University of Göttingen (Other); Esbjerg Hospital - University Hospital of Southern Denmark (Other); University Hospital Heidelberg (Other); AZ Monica Campus Antwerpen (Unknown); Academisch Ziekenhuis Maastricht (Other); Radboud University Medical Center (Other)
Responsible Party: Principal Investigator, Gwen Swennen, maxillofacial surgeon, principal investigator, AZ Sint-Jan AV
Other Study IDs: 2004-MC
Record Dates: First submitted 2019-02-14; First posted 2019-02-15 (Actual); Last update posted 2019-06-17 (Actual); Status verified 2019-06

CONDITIONS: Orthognathic Surgery
Keywords: 3D virtual planning software; Individual Patient Solutions Case Designer (IPSCD); timing; international; multicenter

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background Three-dimensional (3D) imaging and subsequent 3D virtual treatment planning are becoming state of the art in orthognathic surgery. However, current available software is still too time-consuming. KLS Martin (Tuttlingen, Germany) has currently completed the preclinical and the single surgeon (GS) closed beta-phase of their novel 3D virtual planning software, IPS (Individual Patient Solutions) CaseDesigner (IPSCD).

Objectives The investigators aim to test pre-release versions of the IPSCD software under real-world working conditions in strictly selected university, general and private hospital settings. In specific, they aim to demonstrate that the IPSCD will ensure a significant reduction in treatment planning time.

Study design closed beta-phase; international, multi-centric, prospective study Patients presenting at the division of maxillofacial surgery at the different hospital centers, for an orthognathic-related problem will receive a complete routine work-up, including a cone-beam CT (CBCT) according to the IPSCD protocol. The same surgeon and/or orthodontist will run all the virtual planning steps with the novel software. Timing of the eight major steps will be measured with a digital chronometer.

One hundred and eight patient cases will be planned with the IPSCD software in the participating centers over a period of three months, in the order of respectively one, three and five cases per month per participating center.

Investigators will register anonymized patient demographics (age, gender, clinical diagnosis, type of surgery), and provide feedback regarding the required time to complete the different surgical planning steps, regarding the number of failed alignments, and the occurrence of software bugs. Intergroup comparison of virtual planning time between the different centers will be analyzed. In addition, the learning effect will be examined through comparison of the different cases planned by the same surgeon and/or orthodontist, or in comparison to the initial beta-testing phase results by GS.

ELIGIBILITY:
Inclusion Criteria:

* Patients of all ages
* Patients of both genders
* Patients should present themselves at the division of Maxillofacial surgery or Orthodontics, at the participating hospital centers for orthognathic surgery
* Patients should receive standardized cone-beam computed tomography (CBCT) image acquisition, according to the IPSCD protocol
* Preoperative 3D virtual planning should be performed by the same investigator per center with the IPSCD software

Exclusion Criteria:

* All patients that do not fit the abovementioned description
* Patients with posttraumatic deformity
* Patients with congenital deformity
* Patients with pre-prosthetic indication

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: All consecutive patients who present themselves at the division of Maxillofacial surgery or Orthodontics, at the participating hospital centers for orthognathic surgery between May and August 2016
Sampling Method: Non-Probability Sample
Enrollment: 69 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2016-09-30 (Actual); Study Completion 2017-03-31 (Actual)

PRIMARY OUTCOMES:
required time to complete total 3D virtual planning | preoperative
  required time to complete total 3D virtual planning, measured in seconds with a digital chronometer

SECONDARY OUTCOMES:
required time to complete the 8 major virtual planning steps | preoperative
  required time to complete the 8 major virtual planning steps, measured in seconds with a digital chronometer

CONTACTS AND LOCATIONS:
Overall Officials: Gwen Swennen, Principal Investigator — department of maxillofacial surgery, AZ Sint-Jan Brugge-Oostende AV

IPD SHARING:
Plan to Share IPD: No